CLINICAL TRIAL: NCT03065569
Title: A Comparison of Epidural Techniques for Labour Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Anton Chau, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H16-03380
Record Dates: First submitted 2017-01-19; First posted 2017-02-28 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Labour Analgesia
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Epidural Technique (Active Comparator): Epidural will be performed Initial dose of 16 mL of 0.125% bupivacaine will be given Upon patient request, rescue bolus based on protocol will be administered.
  Interventions: Drug: Bupivacaine
- Combined Spinal Epidural Technique (Experimental): CSE will be performed Initial dose of 16 mL of 0.125% bupivacaine will be given Upon patient request, rescue bolus based on protocol will be administered.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — 16 mL of 0.125% bupivacaine

SUMMARY:
A trial comparing outcomes for different epidural techniques in labour analgesia

DETAILED DESCRIPTION:
Epidurals are the most common form of pain relief in labour. There are two techniques in use at the moment to place the epidural: epidural or combined spinal epidural (CSE). CSE has been shown to work faster and provide better pain relief than epidural alone. The investigators aim to show that CSE also requires less medication over the course of labour as this may mean it has fewer side effects. The amount of medication needed during labour between the two different techniques given in a standardized way will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, singleton presentation at term

Exclusion Criteria:

* Significant comorbidities likely to alter outcome of labour

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-05-07 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Bupivacaine requirement for analgesia | From randomization until delivery
  milligram of bupivacaine used per hour

CONTACTS AND LOCATIONS:
Overall Officials: Anton Chau, MD MMSc, Principal Investigator — UBC
Locations (2):
- Canada (2):
  - BC Women's Hospital, Vancouver, British Columbia
  - British Columbia's Women's Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No